CLINICAL TRIAL: NCT02837939
Title: Prospective Randomized Single-blind Study on Transfer-factor in Acute Decompensation of Advanced Chronic Liver Disease and Acute-on-chronic Liver Failure.
Brief Title: Transfer Factor Efficacy in the Management of Cirrhosis-associated Immune Dysfunction
Acronym: IMUNO-HEGITO7
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Martin Janičko (Other)
Collaborators: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other)
Responsible Party: Sponsor-Investigator, Martin Janičko, Assistant Professor of Medicine, Faculty of Medicine, Pavol Jozef Safarik University
Organization: Pavol Jozef Safarik University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IMUNO - HEGITO 7
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cirrhosis; Liver Failure
MeSH Terms: conditions — Fibrosis; Liver Failure | interventions — Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Drug: Human derived Transfer factor applied by subcutaneous injection in specified time points.
  Interventions: Drug: Human derived Transfer factor
- Control (Placebo Comparator): Aqua pro injectione 4 mL ampules for subcutaneous administration in the same time points as in the active arm
  Interventions: Drug: Aqua pro injectione 4ml ampules for subcutaneous injection

INTERVENTIONS:
Drug: Human derived Transfer factor — One dose (the content of one amp.) of lyophilised drug contains:
  Leucocyte dialysatum 200 x 10 to the power of 6 (Lyophilized dialysate from 200 million leukocytes) pH = 7.8 to 9 after reconstitution (dissolving) of drug
  To be administered subcutaneously as follows:
  12 doses TF in total:
  * 3 x TF in first week: day 1,3,5
  * 2 x TF in week 2: day 8 , 11
  * 1 xTF in week 3 and 4 : day 15, 22
  * 1 x TF once a month up to 6 month
  Other Names: IMMODIN. Holder: IMUNA PHARM a.s. - GRIFOLS (SVK) Registration number: 59/0147/89-CS
  Arms: Active
Drug: Aqua pro injectione 4ml ampules for subcutaneous injection — 12 doses in total:
  * 3 doses in first week: day 1,3,5
  * 2 doses in week 2: day 8 , 11
  * 1 dose in week 3 and 4 : day 15, 22
  * 1 dose once a month up to 6 month
  Arms: Control

SUMMARY:
This study is aimed to assess the efficacy of Human derived Transfer factor ( T-lymphocytes homogenate that contains small molecular weight (10 kDa) molecules: various IFNs, ILs, chemokines, endorfins, heat shock proteins) in decreasing rate and/or severity of infections in acute or chronic decompensations of liver cirrhosis and acute on chronic liver failure..

DETAILED DESCRIPTION:
Most of mortality from advanced chronic liver disease (ACLD) is mediated by so- called specific complications of end-stage liver disease (ESLD); one of the most important is infection (25-30%). Infection is responsible for considerable proportion of ESLD-related mortality. Important in pathogenesis of infections in ESLD is CAIDS (cirrhosis - associated immune dysfunction syndrome), recently re-named to CAID (Cirrhosis-Associated Immune Deficit). TRANSFER FACTOR (TF) is supposed to act at several points in CAID - cascade. This gave rise to hypothesis, that TF could be of benefit in AD/ACLF.

Characteristics of TF It has been shown that transmission fo T-Lymphocyte reactivity is transmissible not only by T-cells alone, but also by hommogenate of peripheral white blood cells. Later it became clear that for the transmission of cellular immunity is responsible dialysable fraction of T-lymphocytes homogenate (with small molecular weight of 10 kDa; consists of amino acids, small peptides, nucleotides etc). This homogenate was named Transfer - factor (TF). One dose of lyophilized drug contains: Leucocyti dialysatum 200 x 10 6 (contains various IFNs, ILs, chemokines, endorfins, heat shock protein etc)

* stimulates T H 1 response
* induces production of IL-1, IL-2
* activates chemotaxis of immunocompetent cells
* increases fagocytic activity
* activates antigen-presentation by APCs

The aim of this study is to assess the efficacy of transfer factor in decreasing rate and/or severity of infections in ACLF.

ELIGIBILITY:
Inclusion Criteria:

* admission to hospital at participating liver units or ICUs or internal medicine wards with acute decompensation (AD) of advanced chronic liver disease or acute-on-chronic liver failure according to CLIF - C criteria
* ability to provide informed consent,

Exclusion Criteria:

* disapproval
* lymphoproliferative disorders
* liver transplantation in the past
* pregnancy
* suspected. chronic infection in risk locations
* CNS
* peritoneum
* Known virus-related immune deficiency
* malignancy
* severe heart failure (NYHA >= III)
* severe lung disease (COPD, GOLD>3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint that includes the incidence specified infections: | Two years
  1. Spontaneous bacterial peritonitis
  2. Urinary tract infections:
  3. Pneumonia
  4. Skin and soft tissue infections
  5. Spontaneous bacteremia
  6. Endocarditis
  7. Tuberculosis
  8. Infectious colitis

SECONDARY OUTCOMES:
Length of hospital stay | Two years
  The length of hospital stay after the admission with diagnosed infection or contraction of infection during hospital stay
The usage of antibiotics required for treatment of a diagnosed infection | Two years
The incidence of adverse effects | 2 years

OTHER OUTCOMES:
Change in the phagocytic activity of macrophages | 6 months
Changes in the levels of imunoglobulins IgA, IgG, IgM, IgD, IgE | 6 months
Changes in the capacity for oxidative burst in macrophages | 6 months
Changes in the complement levels and activation pathways activity | 6 months
Changes in lymphocyte subpopulations | 6 months
Changes in the levels of immunomodulators - IL-6, TNF alpha | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lubomir Skladany, MD, PhD, Principal Investigator — F.D.Roosevelt Teaching Hospital with policlinic, Banska Bystrica, Slovakia, 97517
Locations (1):
- F.D.Roosevelt Teaching Hospital with policlinic Banska Bystrica, Banská Bystrica, Slovakia